CLINICAL TRIAL: NCT06610214
Title: IMPACT-care (Improved Medication Communication and Patient Involvement at Care Transitions)
Acronym: IMPACT-care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University Hospital (Other)
Collaborators: The Kamprad Family Foundation for Entrepreneurship, Research & Charity (Other); Regional Research Council Mid Sweden (Unknown); Uppsala University (Other)
Responsible Party: Principal Investigator, Ulrika Gillespie, Deputy Chief Pharmacist / Associate Professor, Uppsala University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: UppsalaUH1
Record Dates: First submitted 2024-09-05; First posted 2024-09-24 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Continuity of Patient Care
Keywords: aged; pharmacist intervention; health communication; patient centered care; medication safety; medication information; hospital discharge

STUDY DESIGN:
Intervention Model Description: We plan a prospective intervention study primarily with a before-and-after design. A secondary analysis using an Interrupted Time Series (ITS) design will be conducted with an exploratory approach.
Who Masked: Outcomes Assessor
Masking Description: The assessor of the primary outcome measure will be blinded.
  The secondary outcome measure concerning drug related readmissions will be blinded.
  The secondary outcome measure concerning medication adherence is not possible to blind since it is dependent on the patients' discharge date, and the date will reveal the allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): No intervention
- Intervention group (Experimental): IMPACT-care intervention
  Interventions: Other: IMPACT-care intervention

INTERVENTIONS:
Other: IMPACT-care intervention — 1, Information package for patient and/or caregiver; 2, Preparation of medication-related discharge documentation; 3, Facilitation of discharge communication; 4, Post-discharge follow-up call
  Arms: Intervention group

SUMMARY:
Background: Transitions of care, especially at hospital discharge, pose significant risks to patient safety. The World Health Organization (WHO) identifies this as a critical area for improvement, particularly for older patients who frequently experience preventable adverse drug events (ADEs) post-discharge.These risks often stem from poor communication between hospitals and subsequent care providers, and inadequate communication with patients and their informal caregivers, leading to gaps in post-discharge care. In Sweden, discharge conversations between hospital physicians and patients are standard practice but often lack structure and patient-centeredness. This can result in patients being poorly prepared for self-care, especially in managing their medications.

Aim: To improve the discharge process for older patients, making them (and/or informal caregiver) more informed and involved in their overall care, particularly in medication management.

Design: Prospective intervention study with a before-and-after design, supplemented by an Interrupted Time Series (ITS) analysis using an exploratory approach.

Setting: Two surgical and one geriatric ward in Region Uppsala.

Participants: Patients aged 65 or older, managing medication independently or with assistance from an informal caregiver.

Exclusion: Late palliative stage or transition to it during hospital stay; transfer to a non-participating ward; residence outside the hospital's county; admission from or discharge to a nursing home or short-term care facility; inability to receive information and give consent independently (e.g., cognitive impairment, non-contactable); death during hospital stay; inability to communicate in Swedish; previous inclusion in the study; relocation where another department maintains care responsibility; no persistent medication change post-discharge; hospital stay on the study ward of less than 48 weekday hours.

Interventions: 1, Information package for patient and/or informal caregiver 2, Preparation of medication-related discharge documentation; 3, Facilitation of discharge communication; 4, Post-discharge follow-up call

Primary outcome measure: Quality of medication-related discharge documentation.

Data collection and analyses: Data will be collected from patients' electronic health records (EHR), the Swedish National Board of Health and Welfare's Pharmaceutical Register, and research surveys. Analyses will follow the intention-to-treat principle, using descriptive statistics, t-tests for continuous variables, and chi-square tests for categorical variables.

Relevance: The study aims to enhance the quality of discharge documentation, improve patients adherence to medication changes, increase their sense of participation and involvement in their overall care, and reduce healthcare consumption.

DETAILED DESCRIPTION:
Background:

The global older population is increasing, with the percentage of individuals aged 65 and older expected to rise from 10% in 2022 to 16% by 2050. Older people often suffer from multiple illnesses, doubling their risk of requiring hospital care compared to younger adults. Medication is the most common treatment for various health conditions, and the prevalence of multiple illnesses increases medication usage, heightening the risk of medication-related morbidity. Up to one in five hospital admissions among the older patients is estimated to be medication-related, with most deemed avoidable. Transitions in care, particularly when patients are discharged from the hospital, pose a significant risk to patient safety, highlighted as a a focus area for healthcare improvement by the World Health Organization (WHO). Over one-third of older patients experience adverse drug reactions (ADRs) within eight weeks post-discharge, half of which are considered preventable. These risks are often due to poor communication and coordination between hospitals and subsequent care providers, as well as inadequate communication between healthcare providers and patients/informal caregivers, leading to gaps in patient care post-discharge. Most hospitalized older patients undergo changes in their medication regimens that persist after discharge. Follow-up on these medication changes by subsequent healthcare provider relies on timely and high-quality discharge notes and referrals from hospital physicians, which is not always the case. These well-documented communication issues at discharge have also been confirmed in the Uppsala and Västmanland regions.

In Sweden, it is clinical practice for physicians to have a conversation with the patient at discharge discussing what occurred during the hospital stay. However, these conversations often lack standardized structure and patient-centeredness, appearing more as a checklist item for healthcare staff to complete before discharge. Patient-centered communication at discharge is crucial for preparing patients for self-care including medication management. Involving patients in medical decisions can be part of a patient-centered approach that improves patient satisfaction with care and clinical outcomes (e.g., better glycemic control in diabetics and improved blood pressure control in hypertensives). Challenges exist in involving older patients as they may be less willing and/or able to participate in medical decisions, linked to patient factors such as multimorbidity, cognitive impairment, and hearing loss. It is also common for older patients to express a lack of sufficient medication knowledge, trusting healthcare staff and following prescriptions to the best of their ability without further discussion. Additionally, older patients often struggle to remember medication information communicated at discharge, even when it is presented in a structured manner. Physicians also tend to adopt an authoritative role in medication communication with the patients at discharge, which can reduce the older patients' initiative to engage in their care and medication management. For older patients to be involved in their care at discharge, it is important for healthcare staff to see themselves as advocates for the patient rather than adopting a paternalistic approach in their communication. Informal caregivers also play a crucial role in involving the patient and bridging the communication gap between healthcare staff and the older patients.

With this background, the investigators have initiated the research project IMPACT-care (Improved Medication Information and Patient Involvement at Care Transitions; a strengthened chain of medication information across care boundaries). Within the project, the investigators have conducted several sub-studies exploring medication communication, both oral and written, in connection with the discharge of older patients from hospitals. Based on the results from these sub-studies and the literature, the investigators now plan to conduct the following intervention study with the overall aim of improving medication communication in the discharge process for older patients.

Aim:

To improve the discharge process for older patients, making them (and/or informal caregiver) more informed and involved in their overall care, particularly in their medication management.

Primary objectives:

* Improved medication-related discharge communication.
* Increased patient (and informal caregiver) involvement and confidence in their care in general and their medication management in particular.
* Enhanced patient adherence to medication changes made during the hospital stay and that persist post-discharge.
* Reduced unplanned healthcare utilization post-discharge.

Methods:

The study will be conducted in two surgical and one geriatric ward at the Uppsala University hospital in Region Uppsala.

The study will consist of three phases, the control phase, the training phase, and the intervention phase. Patients will be recruited by the research coordinators and the intervention will be performed by existing workforce at the wards. All healthcare staff involved, i.e., doctors, nurses, and clinical pharmacists, will be trained to perform the intervention. Based on a pilot study, the control and intervention phases will last about six months each and the training phase about four months. Follow-up of included patients will continue up to four months after discharge from the hospital.

The intervention comprises for individual intervention components:

1. Information package for the patient and/or informal caregiver:

   An informational brochure, with a medication focus, and a supplementary informational video (3 minutes in length) based on the information in the brochure. The broshure will be translated into additional languages commonly spoken in Sweden and the film will have subtitles in different languages.
2. Preparation of medication-related discharge documentation:

   Documentation of medication changes and follow-up plans in the patients' EHR supporting the writing of the medication report in the discharge letter and discharge summary.
3. Facilitation of discharge communication:

   Prompting the patient/informal caregiver to review the informational brochure and/or video. Answering questions from patient/informal caregiver about the discharge process. Facilitating the involvement of informal caregivers in the discharge conversation.
4. Follow-up call after discharge:

A call to review the information in the discharge letter and the medication list.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 or older
* Manages medication independently or with assistance from a caregiver

Exclusion Criteria:

* In the late palliative phase of care before or during the hospital stay
* Transfer to a non-participating ward
* Residence outside the hospital's county
* Admission from or discharge to a nursing home or short-term care facility
* Inability to independently receive information and give consent independently (e.g., cognitive impairment, non-contactable)
* Death during hospital stay
* Inability to communicate in Swedish
* Previous inclusion in the study
* Relocation where another department maintains care responsibility
* No persistent medication change post-discharge
* Hospital stay on the study ward of fewer than 48 weekday hours (excluding holidays)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 231 (Actual)
Dates: Start 2024-09-16 (Actual); Primary Completion 2026-01-14 (Actual); Study Completion 2026-01-14 (Actual)

PRIMARY OUTCOMES:
CMDD-M (Complete Medication Documentation at Discharge Measure) | On the 1 day of discharge
  Score (0-9 points) on CMDD-M (Complete Medication Documentation at Discharge Measure). The CMDD-M tool is point-based and measures the accuracy and quality of medication reports in the discharge letter provided to the patient and in the discharge summary intended for the next health care provider. The medication-related discharge documentation is classified as complete if 9 points are achieved using the tool.

SECONDARY OUTCOMES:
PIMCH-Q (Patient Involvement in Medication Communication at Hospital discharge Questionnaire) | Two weeks post discharge
  Score on PIMCH-Q, a questionnaire developed by the research group, administered to patients after discharge, measuring their sense of involvement in medication communication during hospitalization and their sense of knowledge and security related to their medication treatment.
Quality of medication-related discharge documentation | On the 1 day of discharge
  Prevalence of patients with maximum score (9 points) on CMDD-M (patients assessed to have complete medication-related discharge documentation).
Adherence to medication changes made during hospitalization that persist post-discharge, checklist. | Four months post discharge
  - Prevalence of patients without any medication errors
Adherence to medication changes made during hospitalisation that persist post-discharge | Four months post discharge
  - Number of specific medication errors related to lasting medication changes.
Healthcare consumption | 7, 30 and 90 days post-discharge
  - The prevalence of the first unplanned hospital revisit (composite measure of unplanned readmissions and emergency department visits).
Healthcare consumption | 7, 30, and 90 days post-discharge
  - The prevalence of the first unplanned readmission.
Healthcare consumption | 7, 30, and 90 days post-discharge
  - The prevalence of the first emergency department visit (visit not followed by admission).
Healthcare consumption | 7, 30, and 90 days post-discharge
  - The time to the first unplanned hospital revisit.
Healthcare consumption | 7, 30, and 90 days post-discharge
  - The time to the first unplanned readmission.
Healthcare consumption | 7, 30, and 90 days post-discharge
  - The time to the first emergency department visit.
Healthcare consumption | 7, 30, and 90 days post-discharge
  The prevalence of medication-related readmissions. The assessment of whether hospital revisits are medication-related will be conducted using the AT-HARM10 tool.
Healthcare consumption | 7, 30, and 90 days post-discharge
  - The number of unplanned contacts with hospital wards, hospital outpatient clinics, the patient's primary care centre, and the mobile care team.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrika Gillespie, PhD, Principal Investigator — Uppsala University Hospital
Locations (1):
- Uppsala University Hospital, Uppsala, Uppland, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Plan to share individual participant data: Pseudonymised individual participant data from this trial will be made available to researchers upon reasonable request, excluding any direct identifiers. The shared dataset will include all variables relevant to the study findings. Data will be available after publication and for a period of 10 years. Access will be granted to researchers who submit a methodologically sound proposal and agree to use the data solely for scientific purposes, subject to approval by the research team and a data sharing agreement. Requests should be directed to the principal investigator.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: From publication and 10 years forward.
Access Criteria: Access will be granted to researchers who submit a methodologically sound proposal and agree to use the data solely for scientific purposes, subject to approval by the research team and a data sharing agreement. Requests should be directed to the principal investigator.

REFERENCES:
- [Derived] Cam H, Franzon K, Ostman V, Kalvemark Sporrong S, Kempen TGH, Nielsen EI, Lindner KJ, Ekelo B, Bernsten C, Ehlin U, Lindmark S, Hadziosmanovic N, Gillespie U. Improved Medication communication and Patient involvement At Care Transitions (IMPACT-care): study protocol for a pre-post intervention trial in older hospitalised patients. BMJ Open. 2025 May 2;15(5):e099547. doi: 10.1136/bmjopen-2025-099547. PMID 40316362